CLINICAL TRIAL: NCT02155712
Title: Triathlon Tritanium Knee Outcomes Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the pandemic, multiple sites were unable to complete patient visits resulting in less-than-optimal postoperative follow-up occurred. Therefore, study objectives were not met and the decision was made to close the study early.
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Triathlon Tritanium Knee (Active Comparator): Cases are enrolled in the Cohort 1 (cementless) until a total of 356 cases receive the Triathlon Tritanium Tibial Baseplate, Triathlon Tritanium Patella, Triathlon CR or PS Beaded Femur with PA and the Triathlon Tibial Insert. All components in this cohort must used in a cementless application.
  Interventions: Device: Triathlon Tritanium Knee
- Triathlon Knee (Active Comparator): Enrollment in Cohort 2 (cemented) will begin upon completion of enrollment into the Cohort 1 (cementless), and will continue until a total of 144 cases receive the Triathlon Tibial Tray, Triathlon Patella, Triathlon CR or PS Femur and Triathlon Tibial Insert. All components in this cohort must be used in a cemented application.
  Interventions: Device: Triathlon Knee

INTERVENTIONS:
Device: Triathlon Tritanium Knee — Cementless
  Arms: Triathlon Tritanium Knee
Device: Triathlon Knee — Cemented
  Arms: Triathlon Knee

SUMMARY:
The success of the Triathlon Tritanium Knee will be determined by comparing the rate of absence of revision for aseptic loosening of the tibial baseplate at 2 years with the rates reported in the literature.

DETAILED DESCRIPTION:
Cases are to be enrolled at five to ten centers. The same center may be included in both arms. Conversely, a center may choose to participate in only a single arm. The enrollment goal is approximately 36 - 72 cases per center for Cohort 1 (cementless) and 15 - 30 cases per center for Cohort 2 (cemented) , and will vary dependent upon the number of participating centers. Although a goal is presented, there is no maximum limit to the number of cases that a center may enroll. In the event that a center far exceeds the enrollment goal, Stryker may ask the center to cease enrollment so as not to skew the data. All participating centers will comply with the federal regulations regarding patient informed consent and Institutional Review Board (IRB) or Ethics Committee (EC) approval. Non-compliance of a study center may result in termination of the center's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed an Institutional Review Board (IRB)/Ethics Committee (EC) approved; study specific Informed Patient Consent Form.
2. Patient is a male or non-pregnant female age 18-75 years at time of study device implantation.
3. Patient has a diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD).
4. Patient is a candidate for primary cementless total knee replacement, including a resurfaced patella.
5. Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Patient has a Body Mass Index (BMI) > 40.
2. Patient has a diagnosis of avascular necrosis or inflammatory arthritis.
3. Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
4. Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
5. Subject is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.
6. Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
7. Patient is diagnosed with lumbar radicular pain.
8. Patient has a known sensitivity to device materials.
9. Patient is a prisoner.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2023-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Petrow, DO, Principal Investigator — Tucson Orthopaedic Institute; Alvin Ong, MD, Principal Investigator — Rothman Orthopaedic Institute; David Heekin, MD, Principal Investigator — Heekin Clinic; Kipling Sharpe, MD, Principal Investigator — OrthoArizona; Marcus Barnett, MD, Principal Investigator — Mission Hospital Research Institute; John Noble, MD, Principal Investigator — Imperial Health; Michael Masini, MD, Principal Investigator — St. Joseph Mercy Health System; Samuel Wellman, MD, Principal Investigator — Duke University; Ronald Delanois, MD, Principal Investigator — Sinai Hospital of Baltimore; Thomas Bowen, MD, Principal Investigator — Geisinger Orthopaedic Institute
Locations (10):
- United States (10):
  - OrthoArizona, Gilbert, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Heekin Clinic, Jacksonville, Florida
  - Imperial Health, Lake Charles, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - St. Joseph Mercy Health System, Ypsilanti, Michigan
  - Rothman Orthopaedic Institute, Egg Harbor, New Jersey
  - Mission Hospital Research Institute, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Geisinger Orthopaedic Institute, Danville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort 1: 397 participants/451 knees - 78 cases censored leaving 319 participants/373 knees.
  Cohort 2: 216 participants/229 knees - 82 cases censored leaving 134 participants/147 knees.
Groups:
- Cohort 1 Cementless: Cases are enrolled in the Cohort 1 (cementless) until a total of 356 cases receive the Triathlon Tritanium Tibial Baseplate, Triathlon Tritanium Patella, Triathlon CR or PS Beaded Femur with PA and the Triathlon Tibial Insert. All components in this cohort must used in a cementless application.
  It should be noted that Cohort 1 over-enrolled by 17 cases for a total of 373 cases.
- Cohort 2 Cemented: Enrollment in Cohort 2 (cemented) will begin upon completion of enrollment into the Cohort 1 (cementless), and will continue until a total of 144 cases receive the Triathlon Tibial Tray, Triathlon Patella, Triathlon CR or PS Femur and Triathlon Tibial Insert. All components in this cohort must be used in a cemented application.
Period: Overall Study
Arm/Group | Cohort 1 Cementless | Cohort 2 Cemented
Started | 397 | 216
Completed | 0 | 37
Not Completed | 397 | 179
Not completed — Death | 12 | 0
Not completed — Lost to Follow-up | 37 | 22
Not completed — Revision of device | 4 | 3
Not completed — Withdrawal by Subject | 39 | 21
Not completed — Site termination | 77 | 19
Not completed — Sponsor terminated study early | 150 | 0
Not completed — Missed final 5-year protocol visit | 0 | 32
Not completed — Censored because surgery cancelled | 6 | 10
Not completed — Censored because study device was not implanted | 61 | 66
Not completed — Censored because of inclusion/exclusion violation | 11 | 6

BASELINE CHARACTERISTICS:
Population: Includes all participants who received the Triathlon Knee System and were not censored from analysis.
Units Other Than Participants: Knees
Groups:
- Cohort 1 Cementless: Cases are enrolled in the Cohort 1 (cementless) until a total of 356 cases receive the Triathlon Tritanium Tibial Baseplate, Triathlon Tritanium Patella, Triathlon CR or PS Beaded Femur with PA and the Triathlon Tibial Insert. All components in this cohort must used in a cementless application.
  Triathlon Tritanium Knee: Cementless
- Cohort 2 Cemented: Enrollment in Cohort 2 (cemented) will begin upon completion of enrollment into the Cohort 1 (cementless), and will continue until a total of 144 cases receive the Triathlon Tibial Tray, Triathlon Patella, Triathlon CR or PS Femur and Triathlon Tibial Insert. All components in this cohort must be used in a cemented application.
  Triathlon Knee: Cemented
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Cementless | Cohort 2 Cemented | Total
Number analyzed (Participants) | 319 | 134 | 453
Number analyzed (Knees) | 373 | 147 | 520
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.12 (7.19) | 63.18 (7.71) | 62.42 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 57 | 212
  Male | 164 | 77 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 9
  Not Hispanic or Latino | 299 | 127 | 426
  Unknown or Not Reported | 12 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 319 | 134 | 453

OUTCOME MEASURES:

1. Primary Outcome: Number of Knees With Cementless Application That Had Successful Primary Total Knee Replacement With the Triathlon Tritanium Total Knee System
Description: Success is defined as freedom from Triathlon Tritanium Tibial Baseplate revision for aseptic loosening.
Time Frame: 2 years
Population: The primary objective analysis only includes cementless, Cohort 1 participants. All Cohort 2 participants received cemented primary total knee replacements and are not included in the primary objective analysis.
Measure: Number; unit: Successful Knees
Units Other Than Participants: Knees
Groups:
- Cohort 1 Cementless: Cases are enrolled in the Cohort 1 (cementless) until a total of 356 cases receive the Triathlon Tritanium Tibial Baseplate, Triathlon Tritanium Patella, Triathlon CR or PS Beaded Femur with PA and the Triathlon Tibial Insert. All components in this cohort must used in a cementless application.
Arm/Group | Cohort 1 Cementless | Cohort 2 Cemented
Number analyzed (Participants) | 319 | 0
Number analyzed (Knees) | 373 | 0
Successful Knees | 373 |

2. Secondary Outcome: Implant Survivorship (Baseplate and Patella)
Description: This secondary outcome measure is a statistical estimation on the number of cases at risk at 1-year, 3-years, 5-years and 7-years postoperative in the cementless cohort 1 only, per protocol. The final 10-year results were not done due to early study termination.
Time Frame: 10 years
Population: Results below are for the participants/knees that were measured and analyzed at 1-year, 3-year, 5-year, 7-year postoperative on Cohort 1 cementless only as per protocol. The final 10 year was not analyzed due to early study termination.
Measure: Number (95% Confidence Interval); unit: percentage of cementless knees
Units Other Than Participants: Knees
Groups:
- Cohort 1 Cementless: Subjects enrolled in the Cohort 1 (cementless) eligible to receive the Triathlon Tritanium Tibial Baseplate, Triathlon Tritanium Patella, Triathlon CR or PS Beaded Femur with PA and the Triathlon Tibial Insert. All components in this cohort must used in a cementless application.
  Triathlon Tritanium Knee: Cementless
- Cohort 2 Cemented: Subjects enrolled in Cohort 2 (cemented) that began upon completion of Cohort 1 (cementless) enrollment, that were eligible to receive the Triathlon Tibial Tray, Triathlon Patella, Triathlon CR or PS Femur and Triathlon Tibial Insert. All components in this cohort must be used in a cemented application.
  Triathlon Knee: Cemented
Arm/Group | Cohort 1 Cementless | Cohort 2 Cemented
Number analyzed (Participants) | 319 | 0
Number analyzed (Knees) | 373 | 0
percentage of cementless knees
  1-year KM survival rate | 99.42 [97.71 to 99.86] |
  3-year KM survival rate: number analyzed (Participants) | 278 | 0
  3-year KM survival rate: number analyzed (Knees) | 326 | 0
  3-year KM survival rate | 98.74 [96.67 to 99.53] |
  5-year KM survival rate: number analyzed (Participants) | 220 | 0
  5-year KM survival rate: number analyzed (Knees) | 260 | 0
  5-year KM survival rate | 98.74 [96.67 to 99.53] |
  7-year KM survival rate: number analyzed (Participants) | 155 | 0
  7-year KM survival rate: number analyzed (Knees) | 182 | 0
  7-year KM survival rate | 98.05 [95.06 to 99.24] |

3. Secondary Outcome: Compare 2011 Knee Society Score (KSS) Scores Between Both Groups
Description: The 2011 Knee Society Score System is comprised of 4 distinct sub-scores: Objective, Functional, Patient Satisfaction and Expectations. The Objective and Functional sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. The Patient Satisfaction sub-score ranges from a potential minimum score of 0 to a maximum score of 40 points. The Subject Expectations sub-score ranges from a potential minimum score of 0 to a maximum score of 15 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: 2 years
Population: Participants with available data at 2 years are presented for both cohorts.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Cohort 1 Cementless | Cohort 2 Cemented
Number analyzed (Participants) | 244 | 91
Number analyzed (Knees) | 289 | 100
units on a scale
  Objective Knee Score | 94.90 (6.48) | 91.75 (9.40)
  Function Score KSS | 80.85 (15.56) | 75.41 (18.81)
  Patient Satisfaction Score | 35.29 (6.76) | 33.08 (8.06)
  Patient Expectation Score | 10.60 (3.04) | 10.06 (2.89)

4. Secondary Outcome: Compare Oxford Knee Score (OKS) Scores Between Both Groups
Description: The OKS questionnaire consists of 12 questions that cover function and pain of the knee. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes.
Time Frame: 2 years
Population: Participants with available data at 2 years are presented for both cohorts.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Cohort 1 Cementless | Cohort 2 Cemented
Number analyzed (Participants) | 246 | 91
Number analyzed (Knees) | 291 | 100
units on a scale | 42.59 (5.91) | 40.66 (7.79)

5. Secondary Outcome: Compare Short Form-12 (SF-12) Scores Between Both Groups
Description: The SF-12 Health Survey is a 12-item patient quality-of-life questionnaire to measure general health and well-being. It is comprised of two distinct scores (physical and mental component score). They are both calculated on a scale ranging from 0 points to 100 points, with low values representing a poor health state and high values representing a good health state.
Time Frame: 2 years
Population: Participants with available data at 2 years are presented for both cohorts.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Cohort 1 Cementless | Cohort 2 Cemented
Number analyzed (Participants) | 243 | 91
Number analyzed (Knees) | 285 | 100
units on a scale
  SF-12 Physical Component Score | 49.07 (8.36) | 46.24 (9.37)
  SF-12 Mental Component Score | 56.10 (7.46) | 54.28 (8.64)

ADVERSE EVENTS:
Time Frame: Adverse event data is provided from enrollment through the 8-year postoperative interval for the cementless Cohort 1 with a mean of 4.4 years. For the cemented Cohort 2, the period was from enrollment to the 5.6 years postoperative interval with a mean of 3.1 years.
Description: All operative site events occurring at any time, as well as all serious adverse events (SAEs) occurring in the perioperative period (intraoperative to hospital discharge), are collected. Specific Adverse Event terms are not used for all Adverse Events.
Arm/Group | Cohort 1 Cementless | Cohort 2 Cemented
All-Cause Mortality (participants affected / at risk) | 12/319 | 0/134
Serious Adverse Events (participants affected / at risk) | 28/319 | 8/134
Other Adverse Events (participants affected / at risk) | 69/319 | 12/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Cementless (N=319) | Cohort 2 Cemented (N=134)
Non-operative (Cardiac disorders) | 1 (1) | 1 (1)
Non-operative (Gastrointestinal disorders) | 2 (2) | 0 (0)
Operative site (Infections and infestations) | 4 (4) | 1 (1)
Operative site (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Operative site (Musculoskeletal and connective tissue disorders) | 11 (11) | 4 (4)
Non-operative (Nervous system disorders) | 2 (2) | 1 (1)
Non-operative (Renal and urinary disorders) | 3 (3) | 0 (0)
Operative site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Operative site (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Cementless (N=319) | Cohort 2 Cemented (N=134)
Operative site (Musculoskeletal and connective tissue disorders) | 69 (89) | 12 (16) — Events include arthrofibrosis, excessive knee pain, patellar fracture, soft tissue trauma, superficial wound infection, wound hematoma, tendinitis, IT band syndrome, effusion, swelling, bursitis, neuroma, lesion, bruising, incision dehiscence, etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study.These manuscripts & abstracts will be delayed until after the multi-center publication is submitted.All publications shall be submitted to the sponsor for review at least 60 days prior to the submission for publication.The sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-01-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT02155712/Prot_SAP_ICF_000.pdf